CLINICAL TRIAL: NCT06132503
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Clinical Activity of Intravenously Administered LP-284 in Adult Patients With Relapsed or Refractory Lymphomas and Solid Tumors
Brief Title: Safety, Pharmacokinetics, and Clinical Activity of LP-284 in Adult Patients With Relapsed or Refractory Lymphomas and Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lantern Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LP-284-001
Record Dates: First submitted 2023-11-03; First posted 2023-11-15 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Relapsed or Refractory Lymphomas; Advanced Solid Tumor
Keywords: LP-284; Phase 1a/1b; Lantern Pharma; Cancer; lymphoma; DLBCL; MCL; Sarcoma
MeSH Terms: conditions — Recurrence; Lymphoma; Neoplasms; Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase 1 Single Arm Multicenter Study to Assess the Safety and Tolerability of LP-284 (Experimental): The Phase 1a dose escalation portion of the study will identify the maximum tolerated dose (MTD) and/or optimal dose(s) of LP-284 as the RP2D, based on all available safety, PK, PD, and/or preliminary efficacy data. Phase 1b will consist of the dose expansion portion in a separate cohort(s) of patients to further evaluate the safety of LP-284 at the RP2D and obtain preliminary estimates of clinical activity of LP-284 in patients with DLBCL and MCL.
  Interventions: Drug: LP-284

INTERVENTIONS:
Drug: LP-284 — LP-284 is a small molecule alkylating agent causing tumor cell death through DNA damage.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of escalating doses of LP-284 and to determine the maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) in patients with relapsed or refractory (R/R) lymphomas and solid tumors. The secondary objectives are to characterize the pharmacokinetics (PK) of LP-284 and to assess clinical activity of LP-284.

DETAILED DESCRIPTION:
This FIH study is an open-label Phase 1a/1b dose escalation and dose expansion study in adult patients with R/R lymphoma and solid tumors. Patients who provide informed consent and meet the eligibility criteria for the study will be enrolled and treated with LP-284 administered intravenously (IV) on Days 1, 8, 15 of a 28-day schedule.

The study will be conducted in 2 parts: dose escalation with MTD and/or RP2D confirmation (Phase 1a) and dose expansion (Phase 1b). Up to 30 evaluable patients will be enrolled in Phase 1a; the total number of patients will depend on the number of dose levels explored. Up to 40 evaluable patients will be enrolled in each of the 2 cohorts of MCL and DLBCL tumors in Phase 1b.

Patients will remain on study treatment for up to a total of one-year OR until disease progression, unacceptable toxicity, withdrawal of consent, any study-specific discontinuation criteria are met, or the Investigator determines that it is in the best interest of the patient to discontinue study treatment, whichever is shorter.

ELIGIBILITY:
Inclusion Criteria All Patients: Phase 1a and Phase 1b

1. Male or female aged ≥ 18 years on the day of signing informed consent.
2. Patient is capable of giving signed informed consent as described in Section 11.3 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
3. Eastern Cooperative Oncology Group (ECOG) performance status: 0-2 at screening.
4. For Lymphoma patients. At least one bi-dimensionally measurable disease site. The lesion must have a greatest transverse diameter of at least 1.5 cm and greatest perpendicular diameter of at least 1.0 cm at baseline. The lesion must be positive on positron emission tomography (PET) scan.

   Note: Patients without measurable disease per Lugano Classification [9] may be eligible for Part 1a, following discussion with the Investigator and the Sponsor, if the patient presents with non-measurable but assessable disease of any size unequivocally attributable to advanced lymphoma.
5. Adequate organ function at Screening and on C1D1 (pre-dose) defined as:

   Liver Function i Aspartate aminotransferase (AST), alanine transaminase (ALT) ≤ 3x upper limit of normal (ULN) or < 5x ULN in cases of documented lymphoma involvement of liver.

   ii Total serum bilirubin ≤ 1.5 x ULN or < 5x ULN if secondary to Gilbert's syndrome or documented lymphoma involvement of liver.

   Renal Function iii Serum creatinine clearance ≥60 mL/min, either measured or calculated using standard Cockcroft-Gault formula.

   iv Serum electrolyte (potassium, calcium, and magnesium) levels within the normal reference range (may be supplemented according to institutional standards).

   Bone Marrow Function:

   v Absolute neutrophil count (ANC) ≥ 1500/μL. (Phase 1b: ANC ≥ 1000/μL if documented by investigator as the normal baseline for the patient) vi Hemoglobin ≥ 8 g/dL (for those patients undergoing red blood cell [RBC] transfusion, hemoglobin must be evaluated after at least 14 days after the last RBC transfusion).

   vii Platelet count ≥ 100,000/μL (assessed ≥ 7 days following last platelet transfusion in patients with thrombocytopenia requiring platelets). (Phase 1b: ≥ 75,000/μL may be acceptable after discussion with the Sponsor)
6. Women of child-bearing potential (WOCBP) must agree to use highly effective contraceptive methods and avoid egg donation for the duration of study treatment and for 6 months after the last dose of study drug.
7. Women of child-bearing potential must have a negative serum pregnancy test at Screening and within 72 hours prior to the first dose of study drug.
8. Men must agree to use highly effective contraceptive methods and avoid sperm donation during the study treatment and for 3 months after the last dose of study drug if the partner is a WOCBP.

   Phase 1a ONLY:
9. Histologically confirmed diagnosis of B-cell NHL according to the 2016 World Health Organization (WHO) classification that has relapsed from or is refractory to at least two prior standard of care treatments or tumors for whom standard therapies are not available. Diffuse large B-cell lymphoma (DLBCL) includes: DLBCL not otherwise specified (NOS) with or without MYC and BCL2 and/or BCL6 rearrangements; Epstein-Barr virus (EBV) positive DLBCL, NOS; human herpesvirus 8 (HHV8) positive DLBCL, NOS; DLBCL associated with chronic inflammation; and Primary cutaneous DLBCL, leg type. Patients with indolent lymphoma are eligible if they meet criteria for systemic treatment.

   OR Histologically or pathologically confirmed advanced solid tumor that has relapsed from or is refractory to standard treatment, or for which no standard treatment is available.

   Notes: Archival formalin fixed paraffin embedded (FFPE) tumor tissue is preferred but optional.

   Patients with small lymphocytic lymphoma (SLL) are only eligible if they do not require immediate cytoreductive therapy or if they do not have available treatments with potential benefit.

   Patients with solid tumors Only: Non-measurable or Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (Eisenhauer, 2009) for solid tumors at Screening.

   Phase 1b ONLY
10. Histologically confirmed diagnosis of DLBCL or MCL according to the 2016 WHO classification. DLBCL includes: DLBCL not otherwise specified (NOS) with or without MYC and BCL2 and/or BCL6 rearrangements; Epstein-Barr virus (EBV) positive DLBCL, NOS; HHV8+ DLBCL, NOS; DLBCL associated with chronic inflammation; and Primary cutaneous DLBCL, leg type
11. Relapsed and/or refractory disease to at least two prior standard of care treatments or tumors for which no standard therapies are available.
12. Documented tumor alteration status. Archival (preferably collected within 6 months prior to first dose [C1D1]) FFPE tumor sample must be submitted for determination of genomic signature by Lantern Pharma's validated laboratory developed test regardless of whether a local test has been performed for enrollment. The FFPE testing results are not required for study entry.

Exclusion Criteria All Patients: Phase 1a and Phase 1b

Patients are excluded from the study if any of the following criteria apply:

1. History or suspicion of central nervous system (CNS) lymphoma or meningeal involvement or central nervous system (CNS) metastases.
2. History of or active concurrent malignancy other than NHL (Phase 1a and Phase 1b) or solid tumor (Phase 1a only) unless the patient has been disease-free for ≥ 2 years. Exceptions to the ≥ 2-year time limit include treated basal cell or localized squamous cell skin carcinoma, localized prostate cancer, or other localized carcinomas such as carcinoma in situ of cervix, breast, or bladder.
3. Clinically significant AEs that have not returned to baseline or ≤Grade 1 based on NCI-CTCAE prior to first dose of study drug, unless approved by the Sponsor. Patients with chronic Grade 2 toxicities may be eligible per the discretion of the investigator and Sponsor (e.g., Grade 2 chemotherapy-induced neuropathy or hypothyroidism from prior immunotherapy treatment)
4. Ongoing unstable cardiovascular function:

   * Symptomatic ischemia, or
   * Uncontrolled clinically significant conduction abnormalities (i.e., ventricular tachycardia on anti-arrhythmia is excluded; 1st degree atrioventricular block or asymptomatic left anterior fascicular block /right bundle branch block will not be excluded), or
   * Congestive heart failure of New York Heart Association Class ≥ III, or
   * Myocardial infarction within 3 months prior to Screening.
5. Congenital long QT syndrome, or a QT interval corrected by Fridericia's formula (QTcF) ≥ 470 ms (average of triplicate ECGs) at Screening and/or on C1D1 (pre-dose) except for a documented bundle branch block or unless secondary to pacemaker. In the case of a documented bundle branch block or a pacemaker, discussion with the Medical Monitor is required prior to enrollment.
6. Thromboembolic or cerebrovascular event (i.e., transient ischemic attacks, cerebrovascular accidents, pulmonary emboli, or clinically significant deep vein thrombosis) ≤ 6 months prior to first dose of study drug.
7. Infection requiring antibiotics, antivirals, or antifungals within 1 week prior to first dose of study drug, unless such infection is adequately controlled (defined as exhibiting no ongoing signs/symptoms related to the infection and with clinical improvement). In the case of prophylactic use of these agents, discussion with the Medical Monitor is required prior to enrollment.
8. Hepatitis B and/or hepatitis C infection (as detected by positive testing for hepatitis B surface antigen [HbsAg] or antibody to hepatitis C virus with confirmatory testing) or known seropositivity for or history of active viral infection with human immunodeficiency virus (HIV).
9. Concurrent medical conditions including psychiatric disorders that in the judgment of the Investigator will interfere with the patient's ability to participate or with achieving the objectives of the study or pose a safety risk.
10. The patient is pregnant or breastfeeding.
11. Prior allogeneic hematopoietic stem cell transplant.
12. Autologous hematopoietic stem cell transplant within 6 months prior to first dose of study drug or patient has progressed within 6 months from the day of stem cell infusion.
13. Radiation treatment within 4 weeks prior to the first dose of study drug, unless the tumor site continues to increase in size after the patient has completed radiotherapy treatment.
14. Major surgery requiring general anesthesia within 4 weeks prior to the first dose of study drug. If a patient required general anesthesia within the prior 4 weeks, consultation with the Medical Monitor is required prior to enrollment.
15. Received live vaccine within 1 month prior to the first dose of study drug.
16. Exposure to investigational or non-investigational anti-cancer therapy within 2 weeks or within at least 5 half-lives (up to a maximum of 4 weeks from any biologics/immunotherapies) prior to the first dose of study drug, whichever is shorter.

    Note: Low dose steroids (oral prednisone or equivalent ≤ 20 mg/day), localized non-CNS radiotherapy, are not criteria for exclusion.
17. Patient has completed a course of SARS-CoV-2 vaccine within 14 days prior to first dose of study drug.
18. Patient is unable or unwilling to comply with all requirements of the study.
19. Patient with dependency on the Sponsor, Investigator or study site.
20. A person that is committed to an institution by official or judicial order.
21. Male patients with partners currently pregnant or male patients able to father children and female patients of childbearing potential who are unwilling or unable to use highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 3 months (male) or 6 months (female) after last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: To evaluate the safety and tolerability of escalating doses of LP-284 | 12 months
  Evaluate the safety and tolerability of escalating doses of LP-284 by measuring the incidence and severity of adverse events (AEs) of escalating doses of LP-284 to determine the maximum tolerated dose (MTD) in patients with relapsed or refractory (R/R) lymphomas and solid tumors
Phase 1a: To determine the maximum tolerated dose (MTD). | 12 months
  Determine the maximum tolerated dose (MTD) of LP-284 by measuring the incidence and severity of adverse events (AEs) graded according to NCI CTCAE 5.0, clinical laboratory, and electrocardiogram (ECG) abnormalities defined as dose-limiting toxicities (DLTs) in patients with relapsed or refractory (R/R) lymphomas and solid tumors
Phase 1a: To determine the recommended Phase 2 dose (RP2D). | 12 months
  Determine the recommended Phase 2 dose (RP2D) of LP-284 by measuring the incidence and severity of adverse events (AEs) graded according to NCI CTCAE 5.0, clinical laboratory, and electrocardiogram (ECG) abnormalities defined as dose-limiting toxicities (DLTs) in patients with relapsed or refractory (R/R) lymphomas and solid tumors
Phase 1b: To obtain preliminary estimates of clinical activity of LP-284 | 5 years
  To obtain preliminary estimates of clinical activity by examining the overall response rate, based on Investigator's assessment as per Lugano criteria, of LP-284 in adult patients with relapsed/refractory MCL and DLBCL

SECONDARY OUTCOMES:
Phase 1a: To characterize the pharmacokinetics (PK) of LP-284 | 1 year
  To characterize PK parameters for LP-284 and metabolite(s) derived from plasma concentrations
Phase 1a: To assess clinical activity of LP-284 | 1 year
  To obtain preliminary estimates of clinical activity by examining overall response rate based on Investigator's assessment as per Lugano Criteria and Duration of Response (DOR) for lymphoma; and to determine ORR (based on Investigator's assessment), complete response (CR), partial response (PR), and DOR for solid tumors .
Phase 1b: To evaluate the safety and tolerability of LP-284 at the recommended Phase 2 dose(s) (RP2D) | 5 years
  Evaluate the safety and tolerability of LP-284 at the RP2D by measuring the incidence and severity of adverse events (AEs) graded according to NCI CTCAE 5.0, and changes in clinical laboratory parameters, vital signs, and electrocardiograms (ECGs) in patients with relapsed or refractory DLBCL and MCL
Phase 1b: To evaluate clinical activity endpoints for LP-284 | 5 years
  To evaluate duration of response (DOR), progression free survival (PFS) and overall survival (OS) in all in patients with relapsed or refractory DLBCL and MCL. DOR is defined as time of initial response until documented tumor progression, death, or last adequate assessment. PFS is defined as time from treatment initiation to tumor progression, death, or last adequate assessment. OS is defined as time from treatment initiation to death from any cause.
Phase 1b: To characterize the pharmacokinetics (PK) of LP-284 | 5 years
  To characterize PK parameters for LP-284 and metabolite(s) derived from plasma concentrations in patients with relapsed or refractory DLBCL and MCL

CONTACTS AND LOCATIONS:
Overall Officials: Reggie Ewesuedo, MD, Study Director — reggie@lanternpharma.com
Locations (4):
- United States (4):
  - Cancer and Blood Specialists Clinic, Los Alamitos, California
  - Florida Cancer Specialists, Lake Mary, Florida
  - SCRI Oncology Partners, Nashville, Tennessee
  - START Mountain Region, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No